CLINICAL TRIAL: NCT01502332
Title: Comparison of Two Protective Mechanical Ventilation Strategies After Cardiac Surgery: Aggressive Versus Moderate Alveolar Recruitment Strategies
Brief Title: Intensive Alveolar Recruitment Protocol After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Alcino Costa Leme, Supervisor of respiratory post-operative care - Incor Heart Institute, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: InCor-OLA
Record Dates: First submitted 2011-12-21; First posted 2011-12-30 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Ventilator Induced Lung Injury; Cardiac Disease; Acute Lung Injury
Keywords: Mechanical ventilation; Open lung approach; Blood gases; Cardiac surgery; Pulmonary complications
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Heart Diseases; Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Alveolar Recruitment (Experimental): Recruitment with opening pressures of 45 cmH2O in the airways.
  Interventions: Other: Intensive Alveolar Recruitment
- Moderate Alveolar Recruitment (Active Comparator): Recruitment with opening pressures of 20 cmH2O in the airways.
  Interventions: Other: Moderate Alveolar Recruitment

INTERVENTIONS:
Other: Intensive Alveolar Recruitment — Recruitment with opening pressures of 45 cmH2O in the airways, followed by ventilation with PEEP = 13 cmH2O, during 4 hours of protective mechanical ventilation with tidal volume (VT) = 6 mL/kg/pbw.
  Arms: Intensive Alveolar Recruitment
Other: Moderate Alveolar Recruitment — Recruitment with opening pressures of 20 cmH2O in the airways, followed by ventilation with PEEP = 8 cmH2O, during 4 hours of protective mechanical ventilation with VT = 6 mL/kg/pbw.
  Arms: Moderate Alveolar Recruitment

SUMMARY:
The purpose of this study was to evaluate prospectively the impact of two protective mechanical ventilation strategies, both using low tidal volume ventilation (6 mL/kg/ibw) after cardiac surgery. The study selected patients presenting signals of deficient gas exchange (PaO2/FIO2 < 250 at a PEEP [positive end expiratory pressure] of 5 cmH2O) in the immediate post-operative period. An aggressive alveolar recruitment protocol applying opening pressures of 45 cmH2O, followed by ventilation with PEEP = 13 cmH2O, was compared to the standard alveolar recruitment protocol of the institution, where an opening pressure of 20 cmH2O in the airways is followed by ventilation with PEEP = 8 cmH2O. After a stabilizing period of four hours of controlled mechanical ventilation, the patients followed the routine weaning protocol and physiotherapy protocol of the institution.

DETAILED DESCRIPTION:
The postoperative period of cardiac surgery is associated with the development of pulmonary complications. Functional residual capacity can be reduced up to 50% and pulmonary volumes may be decreased until three months after surgery.

Lung injury is the result of pulmonary inflammation (activated by cardiopulmonary bypass, the surgical procedure itself and ischemia-reperfusion injury), the adopted mechanical ventilation strategy and a consequence of previous cardiac and/or pulmonary dysfunction.

The use of protective mechanical ventilation strategies with low tidal volumes since the immediate postoperative period, or since the operating room, has been shown to attenuate and prevent lung injury in previous studies selecting with high-risk patients.

A more complex topic, however, has been the proof of the additional benefit of alveolar recruitment maneuvers during the brief period of mechanical ventilation after surgery. While the experimental evidence suggests that the use of an open lung approach could minimize the shearing forces in the lung parenchyma, enhancing the protection afforded by low tidal volume ventilation, innumerous concerns about the hemodynamic side effects, and the possibility of barotrauma have prevented the routine use of intensive alveolar recruitment protocols. Another matter of concern is the net efficacy of a recruitment maneuver applied in the post-operative period, instead of the intra-operative period.

Thus, this study compared the impact of two protective mechanical ventilation strategies, both using low-tidal volume ventilation (6 mL/kg/ibw) after cardiac surgery, in a selective population of patients presenting signals of deficient gas exchange (PaO2/FIO2 < 250 at a PEEP of 5 cmH2O) in the immediate post-operative period. In a previous study at this institution, this subgroup of patients was shown to be at higher risks of postoperative pulmonary complications.

During the short period of controlled mechanical ventilation after the patient arrival from the operating theater, an aggressive alveolar recruitment protocol applying opening pressures of 45 cmH2O, followed by ventilation with PEEP = 13 cmH2O, was compared to the standard alveolar recruitment protocol of the institution, where an opening pressure of 20 cmH2O in the airways is followed by ventilation with PEEP = 8 cmH2O. After an stabilizing period of four hours of controlled mechanical ventilation, the patients followed the routine weaning protocol and physiotherapy protocol of the institution.

Our hypothesis was that the aggressive alveolar recruitment strategy might help in the reversal of collapse created during the surgery and short term mechanical ventilation during anesthesia and patient transportation. Previous studies have shown that this effect may extend to the post-extubation period, impairing lung function for a few days.

Thus, we tested if the effect of an aggressive alveolar recruitment protocol was translated in a better lung compliance, better gas exchange, and fewer pulmonary complications in the post-operative periods (this latter was our primary outcome). Analysis of the length of stay was also scrutinized, consisting in our secondary outcome. All hemodynamic complications was reported, since we also anticipated that events of hemodynamic impairment might be more frequent in the aggressive recruitment arm, eventually obscuring the expected benefits .

ELIGIBILITY:
Inclusion Criteria:

* Immediate postoperative period of myocardial revascularization and/or heart valve surgery (aortic and/or mitral)
* Age > 18 years and < 80 years
* No previous pulmonary disease
* Left ventricular ejection fraction > 35%
* Body mass index < 40 kg/m2
* Oxygen index (PaO2/FiO2) < 250
* Corrected volemic status (negative raising legs mean arterial pressure [MAP] variation < 10%)
* Written inform consent

Exclusion Criteria:

* MAP (mean arterial pressure) < 60 mmHg
* Noradrenaline > 2 micrograms/Kg/min
* Acute arrhythmias
* Blooding associated to hemodynamic instability
* Need of re-surgery and/or mechanical circulatory assistance
* Suspicion of neurological alteration
* Chest tube with persistent air leak

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2011-12; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo BP Amato, PhD, Study Director — University of Sao Paulo
Locations (1):
- Instituto do Coração (Incor) - University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costa Leme A, Hajjar LA, Volpe MS, Fukushima JT, De Santis Santiago RR, Osawa EA, Pinheiro de Almeida J, Gerent AM, Franco RA, Zanetti Feltrim MI, Nozawa E, de Moraes Coimbra VR, de Moraes Ianotti R, Hashizume CS, Kalil Filho R, Auler JO Jr, Jatene FB, Gomes Galas FR, Amato MB. Effect of Intensive vs Moderate Alveolar Recruitment Strategies Added to Lung-Protective Ventilation on Postoperative Pulmonary Complications: A Randomized Clinical Trial. JAMA. 2017 Apr 11;317(14):1422-1432. doi: 10.1001/jama.2017.2297. PMID 28322416

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Alveolar Recruitment: Intensive Alveolar Recruitment ARM: recruitment with opening pressures of 45 cmH2O in the airways, followed by ventilation with PEEP = 13 cmH2O, during 4 hours of protective mechanical ventilation with VT = 6 mL/kg/pbw.
- Moderate Alveolar Recruitment: Moderate alveolar recruitment ARM: recruitment with opening pressures of 20 cmH2O in the airways, followed by ventilation with PEEP = 8 cmH2O, during 4 hours of protective mechanical ventilation with VT = 6 mL/kg/pbw.
Period: Overall Study
Arm/Group | Intensive Alveolar Recruitment | Moderate Alveolar Recruitment
Started | 157 | 163
Completed | 157 | 163
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intensive Alveolar Recruitment: Recruitment with opening pressures of 45 cmH2O in the airways, followed by ventilation with PEEP = 13 cmH2O, during 4 hours of protective mechanical ventilation with VT = 6 mL/kg/pbw.
- Total: Total of all reporting groups
Arm/Group | Intensive Alveolar Recruitment | Moderate Alveolar Recruitment | Total
Number analyzed (Participants) | 157 | 163 | 320
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 200
  >=65 years | 57 | 63 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [56 to 68] | 63 [57 to 70] | 62 [56 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 66 | 125
  Male | 98 | 97 | 195
Region of Enrollment [Number; unit: participants]
  Brazil | 157 | 163 | 320

OUTCOME MEASURES:

1. Primary Outcome: Severity of Pulmonary Complications in the Post-operative Period
Description: Score of pulmonary complications adapted from previous publications, with 5 degrees, where the higher one means death before hospital discharge, degree (4) means the need of mechanical ventilation for more than 48 hours after surgery or after reintubation, degree (3) means pneumonia or intense noninvasive ventilation need, degree (2) means hypoxemia and abnormal lung findings, degree 1 means simple atelectasis and degree (0) means no complication.
  The comparison used this ordinal variable, representing the highest score achieved during the post-operative period. The comparison between arms was made through the Mann-Whitney U test.
  Data shown are percentage of participants with pulmonary complications grade ≥ 3.
Time Frame: Participants were followed for the duration of hospital stay.
Measure: Number; unit: percentage of participants
Arm/Group | Intensive Alveolar Recruitment | Moderate Alveolar Recruitment
Number analyzed (Participants) | 157 | 163
percentage of participants | 15 | 26
Statistical Analysis 1: Comparison: Intensive Alveolar Recruitment vs Moderate Alveolar Recruitment; Test type: Superiority or Other; p = 0.016, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Length of ICU Stay
Description: Days since surgery until ICU discharge, analyzed through Kaplan-Meyer curves (log-Rank test), where the time to event is the time of discharge from the ICU. The censoring was performed at 28 days. Patients dying before leaving the ICU were censored as not discharged from ICU at day 28.
Time Frame: From the day of surgery up to ICU discharge, maximum censoring at day 28 after surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intensive Alveolar Recruitment | Moderate Alveolar Recruitment
Number analyzed (Participants) | 157 | 163
days | 3 [2 to 4] | 3 [2 to 5]
Statistical Analysis 1: Comparison: Intensive Alveolar Recruitment vs Moderate Alveolar Recruitment; Test type: Superiority or Other; p = 0.014, Log Rank

3. Secondary Outcome: Length of Hospital Stay
Description: Days since surgery until Hospital discharge, analyzed through Kaplan-Meyer curves (log-Rank test), where the time to event is the time of discharge from the Hospital. The censoring was performed at 28 days. Patients dying before leaving the Hospital were censored as not discharged from Hospital at day 28.
Time Frame: From the day of surgery up to Hospital discharge, maximum censoring at day 28 after surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intensive Alveolar Recruitment | Moderate Alveolar Recruitment
Number analyzed (Participants) | 157 | 163
days | 8 [7 to 12] | 9 [7 to 14]
Statistical Analysis 1: Comparison: Intensive Alveolar Recruitment vs Moderate Alveolar Recruitment; Test type: Superiority or Other; p = 0.037, Log Rank

4. Secondary Outcome: Incidence of Barotrauma
Description: Confirmed by X-ray. Test with logistic regression
Time Frame: Five days after surgery
Measure: Number; unit: percentage of participants
Arm/Group | Intensive Alveolar Recruitment | Moderate Alveolar Recruitment
Number analyzed (Participants) | 157 | 163
percentage of participants | 0 | 1

5. Secondary Outcome: Hospital Mortality
Description: Deaths occurred during hospital stay, tested with logistic regression.
Time Frame: From the day of surgery up to Hospital discharge or death, with no maximum censoring.
Measure: Number; unit: percentage of participants
Arm/Group | Intensive Alveolar Recruitment | Moderate Alveolar Recruitment
Number analyzed (Participants) | 157 | 163
percentage of participants | 3 | 5
Statistical Analysis 1: Comparison: Intensive Alveolar Recruitment vs Moderate Alveolar Recruitment; Test type: Superiority or Other; p = 0.267, Regression, Logistic

ADVERSE EVENTS:
Groups:
- Intensive Alveolar Recruitment ARM: Mechanical ventilation strategy: Intensive Alveolar Recruitment ARM: recruitment with opening pressures of 45 cmH2O in the airways, followed by ventilation with PEEP = 13 cmH2O, during 4 hours of protective mechanical ventilation with VT = 6 mL/kg/pbw.
- Moderate Alveolar Recruitment ARM: Mechanical ventilation strategy: Moderate alveolar recruitment ARM: recruitment with opening pressures of 20 cmH2O in the airways, followed by ventilation with PEEP = 8 cmH2O, during 4 hours of protective mechanical ventilation with VT = 6 mL/kg/pbw.
Arm/Group | Intensive Alveolar Recruitment ARM | Moderate Alveolar Recruitment ARM
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/163
Other Adverse Events (participants affected / at risk) | 0/157 | 0/163

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No